CLINICAL TRIAL: NCT04959136
Title: Feasibility Study Of Ambulatory Monitoring System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 205399745
Record Dates: First submitted 2021-05-05; First posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Patient Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ambulatory Monitoring Solution (Experimental): The evaluable device (Ambulatory Monitoring Solution and its parts) is a secondary monitoring device and no decisions/diagnosis will be made from these devices.
  Interventions: Device: Ambulatory Monitoring Solution

INTERVENTIONS:
Device: Ambulatory Monitoring Solution — Aim is to evaluate PR; RR; NIBP, cNIBP, SpO2 and arterial blood pressure with investigational Ambulatory Monitoring Solution (AMS)

SUMMARY:
This is a clinical, data collection study conducted at one site. This study will collect open comments, user feedback and parameter raw data to support patient monitoring product development. Subjects participating in this study will be monitored with the site's standard of care primary monitor and the investigational device as the secondary monitor while enrolled in this study. No subject care decisions or diagnoses will be made based on information obtained from the investigational secondary monitor.

DETAILED DESCRIPTION:
This is a pre-market, open label, prospective, non-randomized, data collection clinical research study conducted at one investigational site. This study will collect open comments, user feedback and parameter raw data to support product development. Raw parameter data will be collected from electrocardiogram (ECG), Pulse Rate (PR), respiratory rate (RR), peripheral capillary oxygen saturation (SpO2), non-invasive blood pressure (NIBP), and temperature. Subjects participating in this study will be monitored with the site's standard of care primary monitor and the investigational device as the secondary monitor while enrolled in this study. No subject care decisions or diagnoses will be made based on information obtained from the investigational secondary monitor.

Participation is expected to last no more than 72 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Are able to provide written informed consent or have a legally designated representative provide written informed consent;
2. Are being cared for in a hospital unit and are expected to remain in the unit for the duration of the study procedure; AND
3. Are an adult 18 years or older, or pediatric or neonate subject.

Exclusion Criteria:

1. Are known to be pregnant;
2. Are breastfeeding; OR
3. Are suffering from infections that require isolation.

Ages: 0 Days to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
User feedback | through study completion, average of one day per subject
  This is an early feasibility study intended to elicit user feedback in a hospital setting in order to improve device functionality and further development of the measurement algorithms. User feedback will be collected by open comments field in CRF.
Collection of electronic parameter data | 2 hours up to 3 days
  Electronic device files from patient sensors will be collected for each subject.

SECONDARY OUTCOMES:
Safety information | through study completion and issues resolved, average of one day per subject
  To collect safety information, including type and number of AEs, SAEs, and device issues.

CONTACTS AND LOCATIONS:
Overall Officials: Rita Linko, Principal Investigator — Hospital District of Helsinki and Uusimaa